CLINICAL TRIAL: NCT02506985
Title: XENITH: Rivaroxaban for Pulmonary Embolism Managed With Catheter Directed Thrombolysis
Acronym: XENITH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Susan Smyth (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Susan Smyth, Principle Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0275-F6A
Record Dates: First submitted 2015-06-17; First posted 2015-07-23 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Embolism; Venous Thrombosis
Keywords: Rivaroxaban; CDT (Catheter directed thrombolysis); PE (pulmonary embolism); NETs; factor Xa
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Focal cortical dysplasia of Taylor | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rivaroxaban (Experimental): For the first 3 weeks, patients will receive rivaroxaban 15mg twice-daily; thereafter they will take rivaroxaban 20mg once-daily as per the drug label. Rivaroxaban will be initiated immediately following completion of alterplase infusion, and heparin will be discontinued at the time of rivaroxaban administration.
  Interventions: Drug: rivaroxaban
- heparin-warfarin (Experimental): Unfractioned heparin (UFH), following hospital protocol to achieve a target PTT or enoxaparin, 1.0mg/kg twice-daily, for a minimal duration of treatment of 5 days. Warfarin may be started on the night after CDT. UFH or enoxaparin should continue until the INR is >= 2.0 on two consecutive measurements at least 24 hours apart with an advised overlap with VKA for 4 to 5 days. VKA dosages will be adjusted to maintain the INR within the therapeutic range (target 2.5, range 2.0 - 3.0).
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: rivaroxaban — Immediately following completion of alteplase infusion, patients will receive rivaroxaban 15 mg oral bid for 21 days followed by 20 mg oral daily.
  Other Names: Xarelto
  Arms: rivaroxaban
Drug: warfarin — Immediately following completion of alteplase infusion, patients will continue on unfractionated heparin or low-molecular weight heparin with initiation of warfarin adjusted to INR of 2-3.
  Other Names: Coumadin
  Arms: heparin-warfarin

SUMMARY:
The trial is an open-label, randomized, trial examining novel biomarkers of thrombosis in patients managed with rivaroxaban vs. standard care following treatment of pulmonary embolism (PE) with catheter-guided alteplase. Patients >18 years old who present with PE and are managed with catheter-guided alteplase will be screened for study inclusion. Patient's meeting inclusion/exclusion criteria will undergo informed consent. Immediately following completion of alteplase infusion, patients will be randomized to receipt of rivaroxaban 15 mg oral bid for 21 days followed by 20mg oral daily or continuation on unfractioned heparin or low-molecular weight heparin with initiation of warfarin adjusted to INR of 2-3. Blood samples will be taken within 2 hours of CDT completion prior to receipt of study treatment (study day 1), at 8h-12h, 24h, 48h, 5d (or prior to hospital discharge), and at 30 day follow-up. Clinical endpoints, including bleeding, evidence of thrombosis progression, and death will be tracked during index hospitalization and at follow-up 30 days post-discharge.

DETAILED DESCRIPTION:
Catheter-guided alteplase has a growing role in the management of acute pulmonary embolism (PE). Following a 12-24 hour alteplase infusion (for bilateral or unilateral PE, respectively) patients are routinely managed with therapeutic unfractionated heparin (UFH) as a bridge to chronic warfarin therapy. It is our desire to study the effects of rivaroxaban vs. standard care following catheter-guided alteplase thrombolytic therapy (CDT) in patients with acute pulmonary embolism. Use of rivaroxaban may offer several important advantages compared to standard therapy in this setting. Among these is the potential for rivaroxaban to improve novel biomarkers of thrombosis including inhibition neutrophil extracellular traps (NETs), tissue factor-positive microparticles, and markers of inflammation. Neutrophil release of extracellular DNA may provide a scaffold upon which venous thrombosis propagates. NETs are associated with thrombus organization. Their dissolution may facilitate thrombolysis. Circulating DNA, a surrogate marker for NETs, is elevated 2-3 fold in patients with venous thromboembolism (VTE) and correlates strongly with plasma myeloperoxidase (MPO), an inflammatory marker of neutrophil and monocyte activation. The investigators have previously demonstrated that heparin can trigger MPO release from leukocytes. Thus, it is resonable to speculate that anti-Xa therapy may reduce inflammation, MPO, and NET levels in circulation. Further, the investigators have observed that catheter-directed thrombolysis may increase length of stay (time frame = 8 hours to 30 days following administration of study drugs) and the investigators would also propose treatment with rivaroxaban may balance this by eliminating a "bridging" period.

ELIGIBILITY:
Inclusion Criteria:

* Provisions of informed consent prior to any study specific procedure
* Diagnosis of acute PE
* Evidence of RV strain as defined by one of the following:
* 1. an RV-to-LV diameter ratio>0.9
* 2. elevated troponin
* 3. elevated BNP
* Plan for CDT for PE.

Exclusion Criteria:

* Arterial hypotension and cardiogenic shock at the time of enrollment. Arterial hypotension defined as a systolic arterial pressure <90mm Hg or a drop in systolic arterial pressure of at least 40 mm Hg for at least 15 minutes with tissue hypoperfusion and/or hypoxia)
* Hypersensitivity or other reaction to rivaroxaban
* Other indication for VKA than PE
* Creatinine clearance <30 ml/min
* Significant liver disease (e.g. acute hepatitis, chronic active hepatitis, cirrhosis) or ALT > 3 x ULN
* Life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Smyth, MD PhD, Principal Investigator — University of Kentucky

REFERENCES:
- [Background] Dahlback B. Advances in understanding pathogenic mechanisms of thrombophilic disorders. Blood. 2008 Jul 1;112(1):19-27. doi: 10.1182/blood-2008-01-077909. PMID 18574041
- [Background] Smith SA, Mutch NJ, Baskar D, Rohloff P, Docampo R, Morrissey JH. Polyphosphate modulates blood coagulation and fibrinolysis. Proc Natl Acad Sci U S A. 2006 Jan 24;103(4):903-8. doi: 10.1073/pnas.0507195103. Epub 2006 Jan 12. PMID 16410357
- [Background] Smith SA, Choi SH, Collins JN, Travers RJ, Cooley BC, Morrissey JH. Inhibition of polyphosphate as a novel strategy for preventing thrombosis and inflammation. Blood. 2012 Dec 20;120(26):5103-10. doi: 10.1182/blood-2012-07-444935. Epub 2012 Sep 11. PMID 22968458
- [Background] Lopez JA, Kearon C, Lee AY. Deep venous thrombosis. Hematology Am Soc Hematol Educ Program. 2004:439-56. doi: 10.1182/asheducation-2004.1.439. PMID 15561697
- [Background] Zhou J, May L, Liao P, Gross PL, Weitz JI. Inferior vena cava ligation rapidly induces tissue factor expression and venous thrombosis in rats. Arterioscler Thromb Vasc Biol. 2009 Jun;29(6):863-9. doi: 10.1161/ATVBAHA.109.185678. Epub 2009 Mar 5. PMID 19265029
- [Background] Bugert P, Pabinger I, Stamer K, Vormittag R, Skeate RC, Wahi MM, Panzer S. The risk for thromboembolic disease in lupus anticoagulant patients due to pathways involving P-selectin and CD154. Thromb Haemost. 2007 Apr;97(4):573-80. PMID 17393020
- [Background] von Bruhl ML, Stark K, Steinhart A, Chandraratne S, Konrad I, Lorenz M, Khandoga A, Tirniceriu A, Coletti R, Kollnberger M, Byrne RA, Laitinen I, Walch A, Brill A, Pfeiler S, Manukyan D, Braun S, Lange P, Riegger J, Ware J, Eckart A, Haidari S, Rudelius M, Schulz C, Echtler K, Brinkmann V, Schwaiger M, Preissner KT, Wagner DD, Mackman N, Engelmann B, Massberg S. Monocytes, neutrophils, and platelets cooperate to initiate and propagate venous thrombosis in mice in vivo. J Exp Med. 2012 Apr 9;209(4):819-35. doi: 10.1084/jem.20112322. Epub 2012 Mar 26. PMID 22451716
- [Background] Ramacciotti E, Myers DD Jr, Wrobleski SK, Deatrick KB, Londy FJ, Rectenwald JE, Henke PK, Schaub RG, Wakefield TW. P-selectin/ PSGL-1 inhibitors versus enoxaparin in the resolution of venous thrombosis: a meta-analysis. Thromb Res. 2010 Apr;125(4):e138-42. doi: 10.1016/j.thromres.2009.10.022. Epub 2009 Dec 4. PMID 19962723
- [Background] Fuchs TA, Brill A, Wagner DD. Neutrophil extracellular trap (NET) impact on deep vein thrombosis. Arterioscler Thromb Vasc Biol. 2012 Aug;32(8):1777-83. doi: 10.1161/ATVBAHA.111.242859. Epub 2012 May 31. PMID 22652600
- [Background] Fuchs TA, Brill A, Duerschmied D, Schatzberg D, Monestier M, Myers DD Jr, Wrobleski SK, Wakefield TW, Hartwig JH, Wagner DD. Extracellular DNA traps promote thrombosis. Proc Natl Acad Sci U S A. 2010 Sep 7;107(36):15880-5. doi: 10.1073/pnas.1005743107. Epub 2010 Aug 23. PMID 20798043
- [Background] Brill A, Fuchs TA, Savchenko AS, Thomas GM, Martinod K, De Meyer SF, Bhandari AA, Wagner DD. Neutrophil extracellular traps promote deep vein thrombosis in mice. J Thromb Haemost. 2012 Jan;10(1):136-44. doi: 10.1111/j.1538-7836.2011.04544.x. PMID 22044575
- [Background] Longstaff C, Varju I, Sotonyi P, Szabo L, Krumrey M, Hoell A, Bota A, Varga Z, Komorowicz E, Kolev K. Mechanical stability and fibrinolytic resistance of clots containing fibrin, DNA, and histones. J Biol Chem. 2013 Mar 8;288(10):6946-56. doi: 10.1074/jbc.M112.404301. Epub 2013 Jan 4. PMID 23293023
- [Background] Bain J, Oyler DR, Smyth SS, Macaulay TE. Pathophysiology and pharmacologic treatment of venous thromboembolism. Curr Drug Targets. 2014 Feb;15(2):199-209. doi: 10.2174/13894501113146660226. PMID 24102472
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivaroxaban | Heparin-warfarin
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Heparin-warfarin | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (17.5) | 50.3 (12.5) | 52.8 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Markers of NETosis at 12h Compared to Baseline
Description: Change in Markers of NETosis at 12h Compared to Baseline
Time Frame: 12h
Population: Sponsor terminated this study and withdrew funding prior to sample analysis. Therefore there was no funding to purchase assays to measure the collected samples nor was there enough samples to complete an assay.
Arm/Group | Rivaroxaban | Heparin-warfarin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Markers of NETosis at 24h Compared to Baseline
Description: Values will be reported in comparison to baseline in the two treatment groups.
Time Frame: 24h
Population: as for outcome 1
Arm/Group | Rivaroxaban | Heparin-warfarin
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Markers of NETosis at 48h Compared to Baseline
Description: Values will be reported in comparison to baseline in the two treatment groups.
Time Frame: 48h
Population: as for outcome 1
Arm/Group | Rivaroxaban | Heparin-warfarin
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Markers of NETosis at 5 Days (or Day of Hospital Discharge) Compared to Baseline
Description: Change in Markers of NETosis at 5 days (or day of hospital discharge) Compared to Baseline. Values will be reported in comparison to baseline in the two treatment groups.
Time Frame: 5 days (or day of hospital discharge)
Population: as for outcome 1
Arm/Group | Rivaroxaban | Heparin-warfarin
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change in Markers of NETosis at 30 Days Compared to Baseline
Description: Values will be reported in comparison to baseline in the two treatment groups.
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | Rivaroxaban | Heparin-warfarin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after hospital discharge
Arm/Group | Rivaroxaban | Heparin-warfarin
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No